CLINICAL TRIAL: NCT00074477
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of 50 and 100 Mg-eq of Paliperidone Palmitate in Patients With Schizophrenia
Brief Title: Safety and Efficacy of an Anti-Psychotic in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004357
Record Dates: First submitted 2003-12-12; First posted 2003-12-15 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; R092670; antipsychotic
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: R092670

SUMMARY:
The purpose of this study is to determine the efficacy (how well the drug works), safety, and side effects of paliperidone palmitate injection compared to placebo in the treatment of the symptoms of schizophrenia in adults. The placebo used in this study was a nutritional substance known as 20% Intralipid emulsion given to patients requiring intravenous feedings.

DETAILED DESCRIPTION:
Paliperidone palmitate is an aqueous suspension that releases paliperidone gradually over a period of about 1 month and is under development to provide a sustained and stable level of paliperidone. This is a randomized (patients will be assigned to different treatment groups based solely on chance), double-blind (neither the patient nor the physician will know if placebo or drug is being given and at what dose), placebo-controlled, multicenter study in patients with schizophrenia. The study consists of a screening period (maximum 5 days, including a 3-day washout of psychotropic medications other than antidepressants, if applicable); a 7-day, open-label, oral run-in period; and a 64-day double-blind treatment period. The total duration of the study is approximately 11 weeks. Efficacy will be evaluated during the study using the Positive and Negative Symptom Scale for Schizophrenia (PANSS) and the Clinical Global Impression - Severity (CGI-S) scale. Safety will be evaluated by monitoring adverse events and changes in clinical laboratory results, including prolactin levels; physical examination results; tardive dyskinesia will be rated using the Abnormal Involuntary Movement Scale (AIMS), akathisia will be rated according to the Barnes Akathisia Rating Scale (BARS), extrapyramidal symptoms will be evaluated using the Simpson-Angus Rating Scale (SAS); electrocardiogram (ECG); vital sign measurements; and concomitant therapy. ER OROS paliperidone (6 or 12 mg) or IR paliperidone (2 or 4 mg) oral dosage administered daily for 7 days (Day -7 to -1), followed by i.m. injections of paliperidone palmitate (either 50 mg eq. or 100 mg eq.), or placebo on Days 1, 8, and 36 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia
* for at least 1 year before screening
* meet PANSS score criteria
* must agree to hospitalization for a minimum of 14 days
* body mass index (BMI) <35.0 kilogram (kg)/meter (m)2.

Exclusion Criteria:

* Patients who are involuntarily committed as in-patients
* have a DSM-IV Axis I diagnosis other than schizophrenia
* have a DSM-IV diagnosis of substance dependence within 3 months before screening (nicotine, caffeine dependence, and history of recreational use of marijuana are not exclusionary)
* have a decrease of >/=25% in the PANSS score between screening and predose
* previous lack of response to 2 adequate trials of antipsychotic treatment
* have a significant risk of suicidal, homicidal, or violent ideation or behavior
* have severe gastrointestinal narrowing (pathologic or iatrogenic)
* current presence of any significant or unstable medication condition
* treatment with any protocol disallowed therapies
* clinically significant result from screening laboratory or ECG.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2003-10; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
The change in total PANSS score from the start of the double-blind treatment period to the end of the double-blind treatment period.

SECONDARY OUTCOMES:
Changes from the start of to the end of the double-blind treatment period in CGI-S and in the PANSS subscales for specific symptoms. Incidence of adverse events, labs and ECGs throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Kramer M, Litman R, Hough D, Lane R, Lim P, Liu Y, Eerdekens M. Paliperidone palmitate, a potential long-acting treatment for patients with schizophrenia. Results of a randomized, double-blind, placebo-controlled efficacy and safety study. Int J Neuropsychopharmacol. 2010 Jun;13(5):635-47. doi: 10.1017/S1461145709990988. Epub 2009 Nov 27. PMID 19941696
- See also: Safety and efficacy of two fixed doses of paliperidone palmitate in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1084&filename=CR004357_CSR.pdf